CLINICAL TRIAL: NCT01034930
Title: A 5-year Prospective Randomised Clinical Study on the Efficiency of Three Different Attachment Systems as Retention for Implant-supported Mandibular Overdenture.
Brief Title: Clinical Study on the Efficiency of Three Different Attachment Systems for Implant-supported Mandibular Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia Dent Srl (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Corina Marilena Cristache, Dr Corina Marilena Cristache, DMD, PhD, senior lecturer, Concordia Dent Srl
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 316/03-207-507
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: MANDIBLE; ATROPHYC EDENTULOUS JAW
Keywords: MANDIBLE; IMPLANTS; OVERDENTURE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Retentive Anchors (Active Comparator): 23 patients will receive as retention system for overdentures Retentive Anchors (Straumann).
  Interventions: Procedure: Insertion of dental implants
- Magnets (Active Comparator): 23 patients will receive Magnets (Straumann) as retention system for overdenture.
  Interventions: Procedure: Insertion of dental implants
- Locator System (Active Comparator): 23 patients will receive Locator System (Straumann) as retention for the mandibular overdenture.
  Interventions: Procedure: Insertion of dental implants

INTERVENTIONS:
Procedure: Insertion of dental implants — Each patient will receive 2 screw-type Straumann (Institut Straumann AG, Basel, Switzerland) standard implants Ø4.1 mm, with SLA surface in the canine region of the mandible with an interconnecting line approaching parallelism with the terminal mandibular hinge axis, according to a standard surgical protocol.
  Other Names: Mandibular overdenture metal reinforced will be made.

SUMMARY:
The aim of the investigators study is to compare, in a prospective controlled clinical trial, the Locator® System with two other types of stress-breaking retention (Retentive Anchors and Magnets) for implant supported overdenture in atrophic edentulous mandible, with the use of Straumann Dental Implant System.

DETAILED DESCRIPTION:
The study was divided in two parts - in the first part of the study 46 fully mandibular edentulous patients will be enrolled. The patients will be recruited from the University Hospital of Dentistry and 9 other private practices in Bucharest and surrounding areas.

Selected patients will be informed about the two different treatment options, about the benefit of treatment with an overdenture retained by two endosseous implants and a written informed consent will be obtained from all participants.

Initial examination

At the beginning of the treatment for each patient will be recorded:

* The medical status.
* The dental history, oral and radiographic examination.
* The hygiene status.
* An evaluation of the existing dentures.
* The estimation of dysfunctional problems.

Treatment procedure Each patient will receive 2 screw-type Straumann (Institut Straumann AG, Basel, Switzerland) standard implants Ø4.1 mm, with SLA surface in the canine region of the mandible with an interconnecting line approaching parallelism with the terminal mandibular hinge axis. The implant lengths will be 10mm and 12mm. The choice of implant length will be dictated by the preoperative radiographic assessment of bone height in the canine region and drilling distance with the principal concern achieving primary stability.

The implants will be inserted under local anaesthesia using a surgical template derived from a tooth wax-up. The implants will be placed in a 1-stage non-submerged procedure according to a strict protocol (Weingart D and ten Bruggenkate 2000). Postoperatively, antibiotics for 5 days treatment (Amoxicillin and Clavulanate Potassium or Erytromycin - for patients alergic to Penicillin), analgesics and Clorhexidine 0,12% mouth rinse will be prescribe for 14 days. Patients will not be allowed to wear the mandibular denture during the first two weeks post-operatively.

One, two and four weeks after the surgical procedure, the patients will be recalled for follow-up visits. At the first recall visit, sutures will be removed. At the second visit the lower denture will be adjusted by selective grinding at the implant location, and Protefix® (Queisser Pharma Germany) Adhesive Cushions will be provided for patients. At all recall visits, patients will receive oral hygiene instructions.

At the third follow-up visit the manufacturing of a new maxillary denture (for the full maxillary edentulous patients) and a mandibular over-denture will be initiated.

After 6 weeks healing period implants will be loaded and the patients will be randomly assigne to one of two main groups:

* Group B of 23 patients will receive retentive anchors (Institut Straumann AG, Basel, Switzerland).
* Group M of 23 patients will receive magnets (Titanmagnetics® Institut Straumann AG, Basel, Switzerland ).

Group B will be randomly divided in two subgroups: full lower denture with two gold matrices with variable retention (four lamellae functioning like a spring - 12 patients and full lower denture with two titanium matrices with defined retention (spring with a defined extraction force of 700-1100g - B.2) - 11 patients. A new mandibular overdenture with metal reinforcement will be made.

The two groups of patients will be compared in the second part of the study with 23 patients receiving Locator system abutments (Group L) following same research protocol.

A new mandibular overdenture with metal reinforcement will be made.

The prosthetic procedure will be performed according the recommendations of the producer (Straumann Dental Implant System) for retentive anchors, magnets and Locator System by experienced prosthodontists. The occlusion will be assessed on the articulator and intra-orally to secure a balanced occlusion in centric relation without anterior tooth contact.

ELIGIBILITY:
Inclusion Criteria:

* Complains about the stability of the existing mandibular denture satisfactory from a technical point of view.
* Acceptance of a mandibular over-denture retained by two endosseous implants.
* Patients agree to a 5-year follow-up period.

Exclusion Criteria:

* Insufficient bone volume (height and with) for inserting at least a 10 mm implant (Ø 4,1).
* Angle class II relationship.
* Physical severe consideration that will affect the minimal invasive surgical procedure or constitute a hindrance for a 5-year follow-up.
* History of radiotherapy in the head and neck region.
* History of pre-prosthetic surgery (including bone graft procedures) or previous oral implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-08; Primary Completion 2009-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The following parameters will be assessed for implant survival: - Gingiva-score, Plaque-score, Calculus, Bleeding-score, Probing pocket depth and Implant stability will be measured using Osstell (RFA). | 5 years

SECONDARY OUTCOMES:
Radiographic outcome: Standardised intra-oral radiographs will be made using the long cone technique. Prosthetic maintenance and complications and soft-tissue complications of the denture bearing area will be recorded. | 5 years
Patient satisfaction will be assessed with the aid of questionnaires: initial (with the original denture), after 6 months, 1-year and 5 years. Final costs for each type of retention will be calculated according to all the procedures and complications. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: CORINA MARILENA I CRISTACHE, DMD, PhD, Principal Investigator — Concordia Dent Srl
Locations (1):
- Concordia Dent Clinic, Bucharest, Romania

REFERENCES:
- [Background] Thomason JM, Feine J, Exley C, Moynihan P, Muller F, Naert I, Ellis JS, Barclay C, Butterworth C, Scott B, Lynch C, Stewardson D, Smith P, Welfare R, Hyde P, McAndrew R, Fenlon M, Barclay S, Barker D. Mandibular two implant-supported overdentures as the first choice standard of care for edentulous patients--the York Consensus Statement. Br Dent J. 2009 Aug 22;207(4):185-6. doi: 10.1038/sj.bdj.2009.728. PMID 19696851
- [Background] Meijer HJ, Raghoebar GM, Batenburg RH, Vissink A. Mandibular overdentures supported by two Branemark, IMZ or ITI implants: a ten-year prospective randomized study. J Clin Periodontol. 2009 Sep;36(9):799-806. doi: 10.1111/j.1600-051X.2009.01442.x. Epub 2009 Jun 26. PMID 19563327
- [Background] Meijer HJ, Raghoebar GM, Batenburg RH, Visser A, Vissink A. Mandibular overdentures supported by two or four endosseous implants: a 10-year clinical trial. Clin Oral Implants Res. 2009 Jul;20(7):722-8. doi: 10.1111/j.1600-0501.2009.01710.x. Epub 2009 Mar 27. PMID 19489933
- [Background] Naert I, Alsaadi G, van Steenberghe D, Quirynen M. A 10-year randomized clinical trial on the influence of splinted and unsplinted oral implants retaining mandibular overdentures: peri-implant outcome. Int J Oral Maxillofac Implants. 2004 Sep-Oct;19(5):695-702. PMID 15508985
- [Background] Naert I, Alsaadi G, Quirynen M. Prosthetic aspects and patient satisfaction with two-implant-retained mandibular overdentures: a 10-year randomized clinical study. Int J Prosthodont. 2004 Jul-Aug;17(4):401-10. PMID 15382775
- [Background] Feine JS, Carlsson GE, Awad MA, Chehade A, Duncan WJ, Gizani S, Head T, Lund JP, MacEntee M, Mericske-Stern R, Mojon P, Morais J, Naert I, Payne AG, Penrod J, Stoker GT, Tawse-Smith A, Taylor TD, Thomason JM, Thomson WM, Wismeijer D. The McGill consensus statement on overdentures. Mandibular two-implant overdentures as first choice standard of care for edentulous patients. Montreal, Quebec, May 24-25, 2002. Int J Oral Maxillofac Implants. 2002 Jul-Aug;17(4):601-2. No abstract available. PMID 12182304
- [Background] Boerrigter EM, van Oort RP, Raghoebar GM, Stegenga B, Schoen PJ, Boering G. A controlled clinical trial of implant-retained mandibular overdentures: clinical aspects. J Oral Rehabil. 1997 Mar;24(3):182-90. PMID 9131473
- [Background] van Steenberghe D, Quirynen M, Naert I, Maffei G, Jacobs R. Marginal bone loss around implants retaining hinging mandibular overdentures, at 4-, 8- and 12-years follow-up. J Clin Periodontol. 2001 Jul;28(7):628-33. doi: 10.1034/j.1600-051x.2001.028007628.x. PMID 11422583
- [Background] Cristache CM, Muntianu LA, Burlibasa M, Didilescu AC. Five-year clinical trial using three attachment systems for implant overdentures. Clin Oral Implants Res. 2014 Feb;25(2):e171-8. doi: 10.1111/clr.12086. Epub 2012 Dec 21. PMID 23278517
- [Result] Cristache CM, Ionescu C, Cristache G, Ionescu I, Iliescu AA, Burlibasa M. A 5-year prospective randomised clinical trial on the efficiency of two different attachment systems as retention for implant-supported mandibular overdenture. Radiographic assessment, cost analysis and final evaluation of treatment's success. Metalurgia International vol. XIV (2009)Special Issue nr. 16:27-34.
- [Result] Cristache CM, Ionescu C, Burlibasa M, Cristache G, Iliescu AA, Dumitriu HT. Retentive anchors versus magnets as attachment systems for mandibular overdenture. A 5-year prospective randomised clinical study.Metalurgia International vol. XIV (2009) special issue no.16: 59-64